CLINICAL TRIAL: NCT04904133
Title: The Effect of Regular Consumption of Low/No Calorie Sweeteners on Glycemic Response and Glucagon Like Peptide-1 Secretion in Healthy Adults: A Randomized Controlled Trial
Brief Title: Effects of Low/No Calorie Sweeteners on Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Şaziye Ecem Örkü, Ph.D, Department of Nutrition and Dietetics, Acıbadem University, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 28850; 218S378 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2021-05-14; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Healthy Population; Glucose Tolerance
Keywords: artificial sweeteners; non-nutritive sweeteners; oral glucose tolerance; glucagon-like peptide-1; insulin secretion; satiety peptides

STUDY DESIGN:
Intervention Model Description: Volunteers were randomly divided into 4 groups (saccharin, sucralose, aspartame+acesulfame-K [Asp+Ace-K], control) and asked to drink the LNCS sweetened water once a day for 4-wks. All study groups and concentration of LNCS they consumed written as follows; Saccharin group: 330 mL water + 140 mg saccharine Sucralose group: 330 mL water + 66 mg sucralose Asp+Ace-K group: 330 mL water + 88 mg aspartame and 88 mg acesulfame-K Control group IV: 330 mL water only
Who Masked: Participant, Investigator
Masking Description: Participants were not informed about the study group and also which sweetener they consumed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saccharine Group (Active Comparator): 140 mg saccharin (Hermesetas) dissolved in 330 mL water for 4 weeks.
  Interventions: Other: Low/No Calorie Sweeteners
- Sucralose Group (Active Comparator): 66 mg sucralose (Splenda) dissolved in 330 mL water for 4 weeks.
  Interventions: Other: Low/No Calorie Sweeteners
- Aspartame+Acesulfame-K Group (Active Comparator): 88 mg aspartame+88 mg acesulfame-K (Takita) dissolved in 330 mL water for 4 weeks.
  Interventions: Other: Low/No Calorie Sweeteners
- Control Group (Placebo Comparator): 330 mL water for 4 weeks.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Low/No Calorie Sweeteners — LNCS powdered and then dissolved in water.
  Arms: Aspartame+Acesulfame-K Group; Saccharine Group; Sucralose Group
Other: Placebo Group — Water
  Other Names: Control
  Arms: Control Group

SUMMARY:
This study aims to determine the effects of chronic exposure to some low/no calorie sweeteners (LNCS) on glucose tolerance and glucagon like peptide 1 (GLP-1) release in healthy individuals. LNCS examined in this study are saccharin, sucralose and aspartame+acesulfame-K. The amounts of LNCS given to the participants are kept similar to daily life exposure; far less than the Acceptable Daily Intakes (ADIs) levels proposed by Food and Drug Administration (FDA) or European Food Safety Authority (EFSA).

DETAILED DESCRIPTION:
Excessive sugar consumption has been related to chronic metabolic problems, including obesity, type 2 diabetes, neuroinflammatory diseases, etc. Therefore, it is recommended to decrease added sugar intake below 10% of total energy intake. Low/no calorie sweeteners (LNCS) may seem as a good alternative to added sugars because they provide sweetness without adding calories to the diet. Although they may reduce energy intake and prevent weight gain, studies investigating the short and long term effects of these sweeteners on metabolic profile are controversial. Therefore, there is a need for future studies to shed light on metabolic effects of these compounds in humans.

Some observational and clinical studies show that they may cause insulin resistance and type 2 diabetes. There are possible mechanisms that may explain this relationship. One of these possible mechanisms is interaction with sweet taste receptors (STRs). It has been shown that STRs not only found in oral cavity but also in extra-oral tissues, such as gastrointestinal tract, pancreas, brain, etc. In vitro studies with sucralose, it has been shown that it may activate STRs in L-cells and stimulate GLP-1 release in a similar manner with glucose. However, these results were not confirmed in vivo.

There are at least six different LNCS approved for human use worldwide. However, each of them have different biological fate in terms of absorption, metabolism and excretion characteristics in the body. Therefore, result of a study with one of LNCS cannot be extrapolated for all LNCS; each of them should be studied in well-designed studies.

In this study it is hypothesized that LNCS may activate STRs in intestinal L-cells and alter release of GLP-1; as a result impair glucose tolerance. In acute human studies, these effects are tested and there are controversial results in regard to glucose tolerance or incretin release. However, individuals who want to consume fewer calories or to better control their blood glucose use LNCS in place of sugar for longer period of time. For this reason, we wanted to test the effects of regular use of LNCS on glucose tolerance and incretin release.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Normoglycemic,
* Female,
* 19-45 years old,
* Weight-stable past 3 months

Exclusion Criteria:

* Insulin resistance,
* Type 2 diabetes mellitus,
* Presence of acute/chronic infection,
* Use of medication that may affect glucose metabolism (thiazide diuretics, glucocorticoids, estrogen or beta blockers)
* Chronic alcohol intake,
* Regular consumption of diet soda (more than one can of soda per week)

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
3 Hours Plasma Glucose | 3 hours
  Change from baseline plasma glucose levels at 4 weeks observed. Participants underwent a 3-h oral glucose tolerance test (3-h OGTT) by consuming a 250 mL 75 g glucose solution, and blood samples were collected at 60, 120, 180 min.
3 Hours Plasma Insulin | 3 hours
  Change from baseline insulin levels at 4 weeks observed. Participants underwent a 3-h oral glucose tolerance test (3-h OGTT) by consuming a 250 mL 75 g glucose solution, and blood samples were collected at 60, 120, 180 min.
Glucagon-like peptide-1 (GLP-1) release | Week 4
  Change from baseline fasting GLP-1 levels at 4 weeks observed.

SECONDARY OUTCOMES:
Body Weight | Week 4
  Change from baseline body weight at 4 weeks observed. Participants were weighed on a digital scale (Tanita MC 180) in fasted state. Weights were expressed in kilograms (kg).
Fat Mass | Week 4
  Change from baseline fat mass (kg) at 4 weeks observed. Fat mass was determined by bioelectrical impedance analysis (BIA) method (Tanita MC180).
Fat-Free Mass | Week 4
  Change from baseline fat-free mass (kg) at 4 weeks observed. Fat-free mass was determined by bioelectrical impedance analysis (BIA) method (Tanita MC180).
Total Body Water | Week 4
  Change from baseline total body water (kg) at 4 weeks observed. Total body water was determined by bioelectrical impedance analysis (BIA) method (Tanita MC180).
Body Mass Index (BMI) | Week 4
  Change from baseline BMI at 4 weeks observed. BMI was calculated as weight (in kilograms) divided by the square of height (in meters).
Waist Circumference | Week 4
  Change from baseline waist circumference (in centimeters) at 4 weeks observed.

CONTACTS AND LOCATIONS:
Overall Officials: Saziye E Orku, Dr., Principal Investigator — Acibadem University
Locations (1):
- Acıbadem Dr. Şinasi Can (Kadıköy) Hospital, Istanbul, Anadolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Rogers PJ, Hogenkamp PS, de Graaf C, Higgs S, Lluch A, Ness AR, Penfold C, Perry R, Putz P, Yeomans MR, Mela DJ. Does low-energy sweetener consumption affect energy intake and body weight? A systematic review, including meta-analyses, of the evidence from human and animal studies. Int J Obes (Lond). 2016 Mar;40(3):381-94. doi: 10.1038/ijo.2015.177. Epub 2015 Sep 14. PMID 26365102
- [Background] Miller PE, Perez V. Low-calorie sweeteners and body weight and composition: a meta-analysis of randomized controlled trials and prospective cohort studies. Am J Clin Nutr. 2014 Sep;100(3):765-77. doi: 10.3945/ajcn.113.082826. Epub 2014 Jun 18. PMID 24944060
- [Background] Toews I, Lohner S, Kullenberg de Gaudry D, Sommer H, Meerpohl JJ. Association between intake of non-sugar sweeteners and health outcomes: systematic review and meta-analyses of randomised and non-randomised controlled trials and observational studies. BMJ. 2019 Jan 2;364:k4718. doi: 10.1136/bmj.k4718. PMID 30602577
- [Background] Romo-Romo A, Aguilar-Salinas CA, Brito-Cordova GX, Gomez Diaz RA, Vilchis Valentin D, Almeda-Valdes P. Effects of the Non-Nutritive Sweeteners on Glucose Metabolism and Appetite Regulating Hormones: Systematic Review of Observational Prospective Studies and Clinical Trials. PLoS One. 2016 Aug 18;11(8):e0161264. doi: 10.1371/journal.pone.0161264. eCollection 2016. PMID 27537496
- [Background] Jang HJ, Kokrashvili Z, Theodorakis MJ, Carlson OD, Kim BJ, Zhou J, Kim HH, Xu X, Chan SL, Juhaszova M, Bernier M, Mosinger B, Margolskee RF, Egan JM. Gut-expressed gustducin and taste receptors regulate secretion of glucagon-like peptide-1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15069-74. doi: 10.1073/pnas.0706890104. Epub 2007 Aug 27. PMID 17724330
- [Background] Brown RJ, Rother KI. Non-nutritive sweeteners and their role in the gastrointestinal tract. J Clin Endocrinol Metab. 2012 Aug;97(8):2597-605. doi: 10.1210/jc.2012-1475. Epub 2012 Jun 7. PMID 22679063
- [Background] Nakagawa Y, Nagasawa M, Yamada S, Hara A, Mogami H, Nikolaev VO, Lohse MJ, Shigemura N, Ninomiya Y, Kojima I. Sweet taste receptor expressed in pancreatic beta-cells activates the calcium and cyclic AMP signaling systems and stimulates insulin secretion. PLoS One. 2009;4(4):e5106. doi: 10.1371/journal.pone.0005106. Epub 2009 Apr 8. PMID 19352508
- [Background] Fujita Y, Wideman RD, Speck M, Asadi A, King DS, Webber TD, Haneda M, Kieffer TJ. Incretin release from gut is acutely enhanced by sugar but not by sweeteners in vivo. Am J Physiol Endocrinol Metab. 2009 Mar;296(3):E473-9. doi: 10.1152/ajpendo.90636.2008. Epub 2008 Dec 23. PMID 19106249
- [Background] Sylvetsky AC, Brown RJ, Blau JE, Walter M, Rother KI. Hormonal responses to non-nutritive sweeteners in water and diet soda. Nutr Metab (Lond). 2016 Oct 21;13:71. doi: 10.1186/s12986-016-0129-3. eCollection 2016. PMID 27777606
- [Background] Ma J, Bellon M, Wishart JM, Young R, Blackshaw LA, Jones KL, Horowitz M, Rayner CK. Effect of the artificial sweetener, sucralose, on gastric emptying and incretin hormone release in healthy subjects. Am J Physiol Gastrointest Liver Physiol. 2009 Apr;296(4):G735-9. doi: 10.1152/ajpgi.90708.2008. Epub 2009 Feb 12. PMID 19221011
- [Background] Temizkan S, Deyneli O, Yasar M, Arpa M, Gunes M, Yazici D, Sirikci O, Haklar G, Imeryuz N, Yavuz DG. Sucralose enhances GLP-1 release and lowers blood glucose in the presence of carbohydrate in healthy subjects but not in patients with type 2 diabetes. Eur J Clin Nutr. 2015 Feb;69(2):162-6. doi: 10.1038/ejcn.2014.208. Epub 2014 Oct 1. PMID 25271009
- [Derived] Orku SE, Suyen G, Bas M. The effect of regular consumption of four low- or no-calorie sweeteners on glycemic response in healthy women: A randomized controlled trial. Nutrition. 2023 Feb;106:111885. doi: 10.1016/j.nut.2022.111885. Epub 2022 Nov 1. PMID 36470113